CLINICAL TRIAL: NCT00255307
Title: A Pilot Evaluation of Two Dosing Schedules of American Ginseng Extract in Pediatric Upper Respiratory Tract Infection.
Brief Title: Pilot Evaluation of CVT-E002 in Pediatric Upper Respiratory Tract Infection.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CV Technologies (Industry)
Collaborators: University of Alberta (Other); Capital Health, Canada (Other)
Organization: Afexa Life Sciences Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVT-E002-2005-4
Record Dates: First submitted 2005-11-16; First posted 2005-11-18 (Estimated); Last update posted 2007-06-18 (Estimated); Status verified 2007-06

CONDITIONS: Upper Respiratory Infection
Keywords: cold; flu; respiratory tract infection
MeSH Terms: conditions — Respiratory Tract Infections; Common Cold; Influenza, Human

INTERVENTIONS:
Drug: CVT-E002 ginseng extract

SUMMARY:
This is a randomized double-blind three-arm trial to evaluate two dosages of CVT-E002 against placebo in pediatric upper respiratory tract infections (URTI). It is hypothesized that CVT-E002 use at standard doses reduces the duration of URTI in children aged 3-12 years.

DETAILED DESCRIPTION:
The eligible children, for whom parental consent has been obtained, will be randomized to one of three groups (standard dose, low dose, or placebo). The standard dose group will receive an oral aqueous solution using the standard dose of CVT-E002, adjusted according to the child's weight. The second group will receive an oral aqueous solution with half of the standard dose of CVT-E002, adjusted according to the child's weight, and the third group will receive a placebo as an aqueous solution of starch that does not contain any CVT-E002 or active medication, volume adjusted for the child's weight. Parents will be provided with a 3-day supply of study medication according to the randomization schedule. CVT-E002 will be administered by the parent to the child three times daily for three consecutive days following the onset of a URTI. Severity and duration of URTI will be measured using the reliable and valid Canadian Acute Respiratory Infection Flu Score (CARIFS).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-12 years who present to their pediatrician with in 48 hours of the onset of an acute upper respiratory tract infection.
* signed informed consent form

Exclusion Criteria:

* Children who have had an immunization in 3 months prior to the study
* Children with known hypoglycemia or diabetes
* Children who have a bacterial illness diagnosed at the same visit (e.g. otitis media, pneumonia, etc.) which will be treated with antibiotic therapy
* Children who have a malignancy or who have undergone treatment for a malignancy in the previous three months
* Children with known active liver disease (e.g. hepatitis)
* Known hypersensitivity to ginseng products
* Concurrent treatment with warfarin, digoxin, ginseng products or phenelzine
* Patients with coagulation disorders

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2005-11; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
To establish preliminary estimate of treatment effect of two doses of American ginseng extract, CVT-E002, in reducing severity and duration of URTI in children

SECONDARY OUTCOMES:
To document adverse events related to the short course of American ginseng extract, CVT-E002, in children

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Vohra, MD, Principal Investigator — University of Alberta/Capital Health
Locations (2):
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Misericordia Child Health Clinic, Edmonton, Alberta

REFERENCES:
- [Derived] Vohra S, Johnston BC, Laycock KL, Midodzi WK, Dhunnoo I, Harris E, Baydala L. Safety and tolerability of North American ginseng extract in the treatment of pediatric upper respiratory tract infection: a phase II randomized, controlled trial of 2 dosing schedules. Pediatrics. 2008 Aug;122(2):e402-10. doi: 10.1542/peds.2007-2186. PMID 18676527